CLINICAL TRIAL: NCT01156714
Title: Effects of Exercise and Cognitive Training on Executive Function in Parkinson's Disease
Brief Title: Exercise and Cognitive Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7158-R
Record Dates: First submitted 2010-03-11; First posted 2010-07-05 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Treadmill Training; Exercise; Cognitive Training; Executive Function; Dual Task
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Treadmill Training (Other): Treadmill training with aerobic exercise
  Interventions: Behavioral: Treadmill training with aerobic exercise
- Arm 2: Memory Training (Other): Memory training with computerized memory program
  Interventions: Behavioral: Memory training with computerized memory program
- Arm 3: Treadmill and Memory Training (Other): Combination of treadmill training and computerized memory program
  Interventions: Behavioral: Combination of treadmill training and computerized memory

INTERVENTIONS:
Behavioral: Treadmill training with aerobic exercise — walk on treadmill for aerobic exercise
  Arms: Arm 1: Treadmill Training
Behavioral: Memory training with computerized memory program — memory testing and training on computer program
  Arms: Arm 2: Memory Training
Behavioral: Combination of treadmill training and computerized memory — both exercise and cognitive computer training
  Arms: Arm 3: Treadmill and Memory Training

SUMMARY:
This study compares the effects treadmill exercise, computerized cognitive training, or the combination of the two on executive function, dual-task performance, and performance on several Instrumental Activities of Daily Living (IADLs).

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is recognized as both a motor and nonmotor disorder. Gait and mobility impairments are often associated with a decline of cognitive function, particularly executive function (EF), among other non-motor signs. EF is a broad category of cognitive functions that is generally defined as those processes necessary for purposeful, goal-directed behavior and supervision of ongoing cognitive processes. Deficits in EF are frequently seen early in PD4 and progress with time, often resulting in disruption of daily activities. People with PD are often impaired in real life situations in which more than one activity needs to be performed at a time. Dual tasking (DT) is defined as the performance of two different tasks simultaneously, commonly a gait plus a cognitive task. This study investigates the interaction of motor (gait) and non-motor (cognitive) impairments in PD. Studies of DT suggest that reciprocal interactions exist between gait and mental functions that are fundamental to the performance of daily activities. Therefore, the model of DT encompasses 2 major areas of PD-related impairment in a single outcome measure that is highly correlated with daily function.

Performance on DT generally results in degradation of gait and/or cognitive performance. The investigators' pilot study in 125 people with PD has shown significant DT interference producing a 22% decline in gait velocity. This demonstrates deterioration of gait performance when subjects allocate attention to the cognitive task. Importantly, deficits on DT correlates with in problems in daily function, especially instrumental activities of daily living (IADLs), and is associated with increased risk of falling and driving impairment. Similarly, the investigators' pilot data in patients with moderate stage PD shows that deficits in DT performance are associated with poor IADL performance. Although cognitive deficits contribute to disability in PD, there are no treatments that effectively address this problem, and no studies have systematically investigated the potential benefits of rehabilitation strategies to improve cognitive function and related disability in this population.

Emerging evidence suggests the potential of physical exercise and cognitive training to improve cognitive function in healthy elderly and individuals with chronic neurologic conditions. A Cochrane meta-analysis on the cognitive effects of aerobic exercise in older adults has shown that improvement of peak VO2 levels by a mean of 14% (range 5-20%) was associated with improvement in cognitive function, particularly EF domains including speed of motor processing and attention. These are the same EF domains in which deficits commonly occur in PD. Pilot data from the investigators' Baltimore VA study show that the investigators can reproduce similar gains in cardiopulmonary fitness in PD, as reported in the Cochrane review, with a 3-month aerobic exercise program. The investigators' group has also reported improvement of selected EF domains (attention and speed of processing) following 2 months of aerobic exercise in stroke patients12. Cognitive training is another potential rehabilitation modality to improve cognitive function. Recent studies in numerous neurological conditions and healthy older adults show that cognitive training improves cognition, with EF most likely to respond among all cognitive domains.

In this project, the investigators are comparing the effectiveness of a treadmill aerobic exercise program (TAEX) versus a cognitive training program (TCOG) versus the combination of TAEX + TCOG for improving EF, DT performance and IADLs in the investigators' sample of Veterans and others with PD.

The investigators' fundamental hypothesis is that 3 months of combined TAEX+TCOG will be most effective in improving EF, DT performance, and IADLs, compared to either regimen alone.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease stage 1-3 Hoehn and Yahr
* Balance problems

Exclusion Criteria:

* unstable medical illness
* unstable psychiatric illness
* exercising too much on own
* doing computerized memory training on own

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Ivey, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Treadmill Training: Treadmill training with aerobic exercise
  treadmill training: walk on treadmill for aerobic exercise
- Arm 2: Memory Training: Memory training with computerized memory program
  computerized memory training: memory testing and training on computer program
- Arm 3: Treadmill and Memory Training: Combination of treadmill training and computerized memory program
  treadmill training: walk on treadmill for aerobic exercise
  computerized memory training: memory testing and training on computer program
Period: Overall Study
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Started | 20 | 19 | 20
Completed | 11 | 15 | 17
Not Completed | 9 | 4 | 3
Not completed — Withdrawal by Subject | 9 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (11.28) | 73.68 (8.38) | 64.55 (7.07) | 67.00 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 15
  Male | 14 | 14 | 16 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 1 | 9
  White | 15 | 14 | 18 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Hoehn & Yahr Parkinson's Disease Severity Rating [Mean (Standard Deviation); unit: units on a scale] — The Hoehn & Yahr scale measures general staging of Parkinson's disease progression. Classification ranges from 1 to 5, with higher scores indicating greater disability. The range of scale scores acceptable for this study was 1 to 3 (1 = Unilateral involvement only, usually with minimal or no functional impairment, 2 = Bilateral or midline involvement, without impairment of balance, 3= First sign of impaired righting reflexes; patients are physically capable of leading independent lives, and their disability is mild to moderate). This assessment was performed by a movement disorders specialist.
  units on a scale | 2.34 (.41) | 2.42 (.42) | 2.35 (.54) | 2.42 (.55)

OUTCOME MEASURES:

1. Primary Outcome: Dual Task Function #1
Description: Dual task tested functional and cognitive performance while walking and talking simultaneously. Walking spatial and temporal parameters were measured using the Gaitrite 24 foot gaitmat with existing hardware and software for analysis.
  Cycle time refers to the amount of time taken for a participant to complete a single stride. Lower scores indicate better outcomes. The range of scores for Cycle Time is: Pre (0.73-2.47), Post (0.72-1.45).
Time Frame: baseline and 3 months
Population: **Please note that initiation of dual-task testing was delayed by the original PI at the start of this study, such that some early participants were missed. This caused the dual-task outcome category to have lower numbers analyzed than other outcomes.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Number analyzed (Participants) | 8 | 13 | 15
seconds
  Cycle Time- baseline | 1.15 (0.152) | 1.12 (.04) | .987 (.037)
  Cycle Time- 3 months | 1.068 (.0375) | 1.09 (.052) | .951 (.035)

2. Primary Outcome: Dual Task Function #2
Description: Dual task tested functional and cognitive performance while walking and talking simultaneously. Walking spatial and temporal parameters were measured using the Gaitrite 24 foot gaitmat with existing hardware and software for analysis.
  Velocity was calculated by dividing the distance by the time it takes to travel that same distance, with consideration for direction. Higher values represent better outcomes. The range of scores for this study was: Pre (36.4 - 269.4), Post (76.3 - 267.6).
Time Frame: baseline and 3 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Number analyzed (Participants) | 8 | 13 | 15
cm/sec
  Velocity- baseline | 131.194 (19.921) | 116.944 (8.213) | 165.165 (11.179)
  Velocity- 3 months | 134.7 (9.016) | 127.353 (10.177) | 174.581 (12.985)

3. Primary Outcome: Cognitive Function #1
Description: 2-Choice Reaction Time measures patients' ability to shift mental set. One of two stimuli are presented on the screen ("+ "or "*"). Subjects press a specified response button on the keyboard corresponding to the presented stimulus. Units are "Throughput", which reflects efficiency of performance by being based on both accuracy and speed. Throughput represents correct responses/ minute.
Time Frame: baseline and 3 months
Measure: Mean (Standard Error); unit: correct responses/ minute
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Number analyzed (Participants) | 11 | 15 | 17
correct responses/ minute
  Two Choice Reaction- baseline | 89.3535 (6.939) | 93.413 (6.227) | 101.236 (4.588)
  Two Choice Reaction- 3 months | 105.677 (7.278) | 103.4767 (5.497) | 119.6465 (5.117)

4. Primary Outcome: Cognitive Function #2
Description: The Stroop is a measure of selective attention and cognitive flexibility in which the subject must inhibit a preponderant response. Subjects are asked to complete three parts under timed conditions: (1) reading words describing colors written in black-and-white, (2) naming those colors when printed as X's, (3) naming the ink color when words describing the colors are mismatched with the colors (suppressing verbal content). Stroop interference scores from condition 3 are t-scores and higher scores equate with better outcomes.
Time Frame: baseline and 3 months
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Number analyzed (Participants) | 11 | 15 | 17
t-score
  Stroop- baseline | 48.37 (1.278) | 41.74 (2.581) | 48.4 (1.54)
  Stroop- 3 months | 48.9 (1.642) | 47.8 (2.522) | 47.941 (1.93)

5. Primary Outcome: Timed Instrumental Activities of Daily Living (TIADL) Function #1
Description: The Timed IADL involves the timing of performance of 5 tasks that mimic everyday instrumental activities of daily living: 1) finding a telephone number in the telephone directory, 2) counting out correct change from a group of coins, 3) finding then reading the ingredients on a food can label, 4) finding two food items in an array of food items (shopping), 5) finding then reading the directions on a medicine container. For each task there is a 2 minute time limit, with the exception of the telephone number task which has a limit of 3 mins. If the task is not completed within the time limit it is terminated. Error codes are assigned for each task. For the tasks completed with minor errors, a time penalty of 1 SD of those who completed the task is added to the completion time. Higher single item scores mean worse performance.The times for each of the tasks are transformed into Z scores which are then summed to form a composite score. Range for shopping item (0.61- 69.9 sec)
Time Frame: baseline and 3 months
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Number analyzed (Participants) | 11 | 15 | 17
z-score
  Timed IADL's Composite- baseline | 0.131 (0.203) | .234 (.164) | -.2435 (0.080)
  Timed IADL's Composite- 3 months | 0.075 (.370) | .1928 (.13866) | -.34 (0.065)

6. Primary Outcome: Timed Instrumental Activities of Daily Living (TIADL) Function #2
Description: The Timed IADL for Shopping involved finding two food items in an array of food items. The task was timed in seconds and if completed with minor errors, a time penalty was added to the completion time. Higher scores/times meant worse performance. The range for shopping task completion was 0.61 to 69.9 seconds.
Time Frame: baseline and 3 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
Number analyzed (Participants) | 11 | 15 | 17
seconds
  TIADL Shopping- baseline | 7.339 (3.856) | 6.01 (1.62) | 3.213 (1.05)
  TIADL Shopping- 3 months | 3.493 (0.980) | 4.746 (1.346) | 2.39 (0.591)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during a 5 month subject participation period which included 1 month of baseline testing, 3 months of intervention, and 1 month of post-testing.
Arm/Group | Arm 1: Treadmill Training | Arm 2: Memory Training | Arm 3: Treadmill and Memory Training
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 1/20
Other Adverse Events (participants affected / at risk) | 5/20 | 3/19 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Treadmill Training (N=20) | Arm 2: Memory Training (N=19) | Arm 3: Treadmill and Memory Training (N=20)
Idiopathic orthostatic hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Participant arrived for study visit and per protocol blood pressure readings were taken which endorsed orthostasis. Participant was taken to ER accompanied by study staff and recovered. Orthostasis is a symptom of PD.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Treadmill Training (N=20) | Arm 2: Memory Training (N=19) | Arm 3: Treadmill and Memory Training (N=20)
fell at home (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (2) | 4 (11) — fall
Grover's disease (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Pt diagnosed during study participation, sought treatment, and was provided prescription topical treatment.
Fell outside at study site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Participant fell outside study site on curb following intervention visit.
migraine headache (General disorders) | 1 (2) | 0 (0) | 1 (1) — participant experienced migraine headache at home.
mild skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — skin irritation from harness used in treadmill training intervention. Participant sought treatment, was given topical ointment, rash cleared.
muscular pain in arm (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) — participant reported arm pain while doing treadmill intervention. Physician assessed participant and suggested he might be holding too tightly to the railing. Participant reported this event on 3 different occasions.
aggravated pre-existing back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) — During treadmill intervention participants reported aggravated back pain.
dystonia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — increase in PD symptom

LIMITATIONS AND CAVEATS:
High drop-out rate across the board, but particularly in Arm 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT01156714/Prot_SAP_000.pdf